CLINICAL TRIAL: NCT06509581
Title: Vitamin E Supplementation for Children With Transfusion Dependent Beta Thalassemia on Different Iron Chelators
Brief Title: Vitamin E Supplementation for Children With Transfusion Dependent Beta Thalassemia on Different Iron Chelation Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amira Abd el moneam, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD12/2020
Record Dates: First submitted 2024-07-06; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Beta-Thalassemia
Keywords: thalasssemia; vitamin E; Oxidative stress
MeSH Terms: conditions — beta-Thalassemia | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta thalassemia patiens with oxidative stress and taking iron chelators receiving vitamin E (Experimental): Beta thalassemia patiens with oxidative stress and taking iron chelators(desferoxamine,deferiprone or deferasirox) receiving vitamin E in dose 400 mg daily for 12 months
  Interventions: Dietary Supplement: vitamin E
- Beta thalassemia patiens with oxidative stress and taking iron chelators receiving placebo (Placebo Comparator): B thalassemia patiens with oxidative stress and taking iron chelators(desferoxamine,deferiprone or deferasirox) receiving placebo for 12 months
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: vitamin E — Vitamin E will be taken for 12 months for beta thalassemia patiens on regular packed red blood cell transfusion and chelators(desferoxamine,deferiprone and deferasirox )
  Arms: Beta thalassemia patiens with oxidative stress and taking iron chelators receiving vitamin E
Other: PLACEBO — placebo will be taken for 12 months for beta thalassemia patiens on regular packed red blood cell transfusion and chelators(desferoxamine,deferiprone and deferasirox )
  Arms: Beta thalassemia patiens with oxidative stress and taking iron chelators receiving placebo

SUMMARY:
repeated transfusions are the mainstay of disease management in most patients with transfusion dependent beta thalassemia.iron overload predispose to oxidative stress and tissue injury.

oxidative stress play important role in pathogenesis of anemia in beta thalassemia.

vitamin E is often depleted in thalassemia patients.

DETAILED DESCRIPTION:
oxidative stress status is very important in thalassemic patients and explains the different manifestations in thalassemic patients.

vitamin E is fat soluble vitamin shown to reduce the oxidative stress in thalassemia and to reduce lipid peroxidation of red cell membranes.

therefore, this study shows the safety of oral vitamin E as adjuvant therapy to three iron chelators : desferoxamine,deferiprone and deferasirox in moderately iron overloaded children and adolescents with transfusion dependent beta thalassemia and its relation to iron overload over one year.

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia patients on regular packed red blood cells transfusion,with vitamin E deficiency
* serum ferritin 1000-2500 ug/l
* cardiacT2*>10ms and ejection fraction >55%

Exclusion Criteria:

* Diabetes,active hepatitis(serum transaminases >2 times ULN)
* renal impairment (serum creatinine>2times ULN)
* participation in previous investigational drug study with 3 months preceding screening supplementation with antioxidants or vitamins within 3 months prior to the study and patients with known allergy to vitamin

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
effect of vitamin E on Liver iron concentration (LIC) | 12 months
  measuring the LIC using MRI (magnetic resonance imaging) in mg/g

SECONDARY OUTCOMES:
effect of vitamin E on antioxidants enzymes | 12 months
  measuring antioxidants enzymes
  * antioxidant enzymes,
effect of vit E supplementation on SF | 12 months
  measuring serum ferritin(SF)in ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fibach E, Rachmilewitz EA. The role of antioxidants and iron chelators in the treatment of oxidative stress in thalassemia. Ann N Y Acad Sci. 2010 Aug;1202:10-6. doi: 10.1111/j.1749-6632.2010.05577.x. PMID 20712766
- [Derived] ElLaboudy MA, Saber MM, Adly AA, Ismail EA, Ibrahim FA, Elalfy OM. Oxidative stress markers and tissue iron overload after 12-months vitamin E supplementation for children with transfusion-dependent beta-thalassemia on different iron chelators: A randomized placebo-controlled trial. Clin Nutr. 2025 Jul;50:154-163. doi: 10.1016/j.clnu.2025.05.003. Epub 2025 May 14. PMID 40424814